CLINICAL TRIAL: NCT04805931
Title: COVID-19 Vaccine Rollout: VEText Message Framing and Covid-19 Vaccine Uptake Among at Risk Veterans
Brief Title: VEText Message Framing and Covid-19 Vaccine Uptake Among at Risk Veterans
Acronym: VEText
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: VA Puget Sound Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Linnaea Schuttner, Staff Physician, VA Puget Sound Health Care System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: COVID-19 Vaccine Rollout
Record Dates: First submitted 2021-03-11; First posted 2021-03-18 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Covid19; Vaccine Refusal
MeSH Terms: conditions — COVID-19; Vaccination Refusal | interventions — Economics, Behavioral

STUDY DESIGN:
Intervention Model Description: Prospective, randomized controlled, parallel groups trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Will receive a text message with standard messaging used to alert veterans that they are eligible for COVID-19 vaccine and offer scheduling embedded within the text message.
- Scarcity (Experimental): Will receive a text message with a behavioral scarcity message used to alert veterans that they are eligible for COVID-19 vaccine and offer scheduling embedded within the text message.
  Interventions: Behavioral: Behavioral economics
- Social good (Experimental): Will receive a text message with a behavioral social good message used to alert veterans that they are eligible for COVID-19 vaccine and offer scheduling embedded within the text message.
  Interventions: Behavioral: Behavioral economics

INTERVENTIONS:
Behavioral: Behavioral economics — Tailored behavioral economic text messaging vs. standard text messaging
  Arms: Scarcity; Social good

SUMMARY:
This is a prospective, randomized controlled trial that will evaluate the effectiveness of two different targeted outreach interventions aimed at increasing Covid-19 vaccine uptake. Veterans who are eligible for COVID-19 vaccine receipt by priority status (based on institutional guidelines) will be identified. Veterans must be enrolled into Veterans Health Administration (VHA) care and meet age or illness institutional priority guidelines to be eligible. Veterans eligible for enrollment into the trial will be randomized in a 1:1:1 allocation at an individual level, using permuted block randomization (with random block sizes of 3 and 6) to the following interventions:

1. Control arm - receives a text message with standard messaging
2. Arm 2 - receives a text message with a message framed for scarcity
3. Arm 3 - receives a text message with a message framed for improving the social good

DETAILED DESCRIPTION:
OBJECTIVE:

To compare the effectiveness of different text message reminders sent through an interactive mobile system (VEText) at increasing Covid-19 vaccine uptake among at risk Veterans.

OVERVIEW:

This is a prospective, randomized controlled trial that will evaluate the effectiveness of two different targeted outreach interventions at increasing Covid-19 vaccine uptake. Veterans who are eligible for Covid-19 vaccine receipt by priority status (based on institutional guidelines) will be identified. Veterans must be enrolled into VHA care and meet age or illness institutional priority guidelines to be eligible. Veterans eligible for enrollment into the trial will be randomized in a 1:1:1 allocation at an individual level, using permuted block randomization (with random block sizes of 3 and 6) to the following interventions:

1. Control arm - receives a text message with standard messaging
2. Arm 2 - receives a text message with a behavioral scarcity message
3. Arm 3 - receives a text message with a behavioral social good message

Randomization will be stratified by VA center (VA Puget Sound or American Lake).

Due to operational constraints, only one type of text message can be sent per day/batch. In order to account for any potential differences with the day of the week the text message is received, the three arm messages will be randomized by day of the week each week. For example, week 1 will have the control group message sent on Monday, the arm 2 message sent on Tuesday, and the arm 3 message sent on Wednesday. Week 2 will have the arm 2 message sent on Monday, the control group message sent on Tuesday, and the arm 3 message sent on Wednesday. Text messages will be sent based on the randomized order generated and will continue on those days of the week that the center has vaccine available.

Our primary outcome of interest is the vaccine scheduling and/or completion rate within 7 days of receipt of the text message. Enrollment in the trial will occur between March 15, 2021 and May 1, 2021.

Primary aims:

Aim 1a: Investigate differences in vaccine scheduling/completion rates among different outreach strategies. Will test the hypothesis (HA1) that the proportion of Veterans either scheduling a vaccine appointment for a first dose or receiving a first vaccine dose varies between targeted behavioral messaging and standard messaging (arms 2 + 3 vs. control) at 7 days post randomization.

Aim 1b: Investigate differences in vaccine scheduling/completion rates among different outreach strategies. Will test the hypothesis (HA1) that the proportion of Veterans either scheduling a vaccine appointment for a first dose or receiving a first vaccine dose varies between different types of behavioral messaging (arm 2 vs. arm 3) at 7 days post randomization.

Secondary aims:

None

Sub-analyses:

None

STUDY POPULATION:

All Veterans who are eligible for a first dose of Covid-19 vaccine by priority status (based on institutional guidelines).

STUDY TIME PERIOD The enrollment period for the study is March 15, 2021 and May 1, 2021. Data collection and analysis will continue through at least 6 months post enrollment for the last Veteran evaluated.

DATA SOURCES:

Table: CDWWork.SVeteran.SMVIPerson Time period: Screening/enrollment Description: Contact information for kit/letter mailing and subsequent reminder calls Variable of interest: Name, address, zip code, phone number, SSN.

Table: CDWWork.SVeteran.SMVIPerson Time period: Screening/enrollment Description: Demographics Analytic variable(s) of interest: DOB, age, gender, marital status, DOD (if applicable), service connectedness, copay.

Table: Communicator report (not CDW table) Time period: Post randomization Description: Provides automated call information Analytic variable(s) of interest: Call date/time, Patient response, Result from non-response.

Table: CDWWork.Appt.Appointment, CDWWork.Dim.Location Time period: Post randomization Description: Scheduled vaccination appointments Analytic variable(s) of interest: Appointment date/time, location.

Table: CDWWork.Immun.Immunization, CDWWork.Dim.ImmunizationName Time period: Post randomization Description: Detailed vaccination receipt records Analytic variable(s) of interest: Vaccine receipt date/time, location.

STATISTICAL ANALYSES AND DESCRIPTION OF MAIN TABLES Sample size analysis assuming a baseline vaccination proportion of approximately 33% among Veterans aged 65 and older (estimates based on vaccination data pulled 03/10/21) the estimated total sample size required to provide at least 80% power to detect a 5% difference between Arms 2 + 3 and the control arm is 4311 total (1437 per group).

Descriptive patient-level statistics will be presented using the Pearson chi-square test for dichotomous variables and the Student's t test for continuous variables. The primary intention-to-treat analysis will use logistic regression to test the association between randomization group and vaccine scheduling/completion 7 days post randomization, adjusting for VHA center as a stratification variable. Odds ratios and predicted probabilities from this model will be reported.

All descriptive and main analyses will be performed using R version 3.6.1. P-values < 0.05 will be considered statistically significant.

1. Aim 1a Statistical Analyses Will test the hypothesis (HA1) that the proportion of Veterans scheduling an appointment for the first vaccine dose or receiving a first vaccine dose varies between targeted behavioral messaging and standard messaging (arms 2 + 3 vs. control) at 7 days post randomization.
2. Aim 1b Statistical Analyses Will test the hypothesis (HA1) that different types of behavioral messaging will have differing effects on vaccine scheduling/vaccine completion at 7 days post randomization (arm 2 vs. arm 3)

STUDY OUTCOMES Primary analyses: % of first-dose vaccine appointments scheduled/vaccines completed at 7 days post randomization

STUDY COVARIATES

Primary analyses:

Covariate of interest: intervention group indicator

ELIGIBILITY:
Eligible participants are automatically enrolled in this project. We are unable to enroll participants upon request.

Inclusion Criteria:

* Veterans must be enrolled into VHA care
* Veterans must meet age or illness institutional priority guidelines for eligibility for COVID-19 vaccine receipt

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4311 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Vaccine appointments scheduled/completed | 7 days post randomization
  % of first-dose vaccine appointments scheduled/vaccines completed

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Reddy, MD, MS, Principal Investigator — VA Puget Sound; Karin Nelson, MD, MSHS, Study Director — VA Puget Sound; Linnaea Schuttner, MD, MD, Principal Investigator — VA Puget Sound; Stefanie Deeds, MD, Principal Investigator — VA Puget Sound
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No